CLINICAL TRIAL: NCT06490445
Title: A Double-blind, Randomized, Placebo-controlled, 4-arm Parallel-group, Multiple-Dose Study to Assess Efficacy and Safety of Medical Cannabis Aerosol Via the Fixed-dose Syqe Inhaler as an Add-on Treatment of Diabetic Peripheral Neuropathic Pain
Brief Title: A Study of Medical Cannabis Aerosol Via the Fixed-dose Syqe Inhaler as an Add-on Treatment of Diabetic Peripheral Neuropathic Pain (DPNP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Syqe Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Syqe-004; 2023-508932-68-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-30; First posted 2024-07-08 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Diabetes; Neuropathy; Painful diabetic neuropathy; Chronic Neuropathic Pain; DPNP; Cannabis; Medical cannabis; Inhaled; Aerosol; Placebo; Randomized; Double-blind
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Marijuana Abuse; Respiratory Aspiration | interventions — Medical Marijuana

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive placebo, inhaled TID via the Fixed-dose Syqe Inhaler.
  Interventions: Drug: Placebo
- 0.25 mg THC (Experimental): Participants will inhale medical cannabis aerosol containing 0.25 mg THC via the Fixed-dose Syqe Inhaler three times a day.
  Interventions: Drug: Medical Cannabis
- 0.5 mg THC (Experimental): Participants will inhale medical cannabis aerosol containing 0.5 mg THC via the Fixed-dose Syqe Inhaler three times a day.
  Interventions: Drug: Medical Cannabis
- 1.0 mg THC (Experimental): Participants will inhale medical cannabis aerosol containing 1.0 mg THC via the Fixed-dose Syqe Inhaler three times a day.
  Interventions: Drug: Medical Cannabis

INTERVENTIONS:
Drug: Medical Cannabis — Syqe cartridge containing medical cannabis (Bedrocan®) administered using Fixed-dose Syqe Inhaler.
  Arms: 0.25 mg THC; 0.5 mg THC; 1.0 mg THC
Drug: Placebo — Placebo administered using Fixed-dose Syqe Inhaler.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of medical cannabis aerosol containing 0.25, 0.5, 1.0 milligrams (mg) delta (Δ)9-tetrahydrocannabinol (THC) inhaled three times a day (TID) compared to placebo via the Fixed-dose Syqe Inhaler on pain intensity at Week 15.

DETAILED DESCRIPTION:
This study will assess the efficacy, safety, tolerability, and pharmacokinetics (PK) of medical cannabis aerosol inhaled via the Syqe Inhaler at nominal doses of 0 (placebo), 0.25, 0.5, and 1.0 mg TID of Δ9-THC added on to standard of care for treatment of DPNP.

The target sample size is 192 eligible participants worldwide, randomized from up to approximately 51 recruiting sites in up to approximately 8 countries.

The study consists of 1) a screening period of up to 14 days; 2) a 15-week, parallel-group, randomized, double-blind treatment period, including a 3-week up-titration period and a 12-week maintenance period; and 3) a post-treatment, safety follow-up period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign the informed consent form (ICF), and willing to abide by the study restrictions.
2. Males and females aged between 18 (included) and 75 (included) years.
3. Agree to use only medical cannabis provided by study team until the end of study (EOS) and not to use any other cannabis or cannabis-containing products.
4. Agree not to participate in other interventional clinical studies during participation in this study.
5. Treated with standard of care for DPNP, either duloxetine or gabapentin or pregabalin as monotherapy or combination of 2.
6. Not current cannabis products users, that is, participants who were previous cannabis products users for any reason but have not used cannabis products within 3 months of the screening visit, or participants who have never used cannabis products, that is, cannabis naïve participants.
7. A diagnosis of DPNP (at screening).
8. Confirmed diagnosis of diabetes mellitus type I or type II with stable disease.
9. Glycated hemoglobin (HbA1c) less than (<) 9% at screening.
10. Body mass index between 18 and 40 kilograms per square meter (kg/m^2), inclusive.
11. Have at least 5 out of 7 records of daily average pain intensity recordings in the 7 days prior to randomization.
12. Agree not to drive or operate heavy machinery during the study treatment period.
13. Female participants must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to the administration of study treatment on Day 1or be of non-child-bearing potential as defined in the protocol.
14. Participants of reproductive potential who are sexually active must use effective birth control methods.

Exclusion Criteria:

1. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol at screening or randomization, ability to complete the study, or study assessments.
2. Presence of skin conditions in the affected dermatome at screening or randomization that could interfere with the evaluation of the neuropathic pain condition.
3. Presence of pain not associated with diabetic peripheral neuropathy (DPN) or other neuropathies that may interfere with study assessments.
4. Known history of significant hypersensitivity, intolerance, adverse reaction or allergy to cannabis products, cannabinoids, or acetaminophen/paracetamol.
5. Malignancies in the past 5 years prior to screening, except for cutaneous basal cell or squamous cell carcinoma resolved by excision.
6. Liver disease or liver injury as indicated by abnormal liver function tests at screening.
7. History or presence of impaired renal function at screening
8. Presence of significant pulmonary disease at screening
9. Ongoing respiratory infection at screening.
10. History of acute coronary syndrome; unstable angina; congestive heart failure; cardiogenic syncope; cardiomyopathy; or symptomatic arrhythmia, or current uncontrolled blood pressure.
11. Concomitant clinically significant cardiac arrhythmias, examples, sustained ventricular tachycardia, and second or third degree atrioventricular block without a pacemaker, or any other relevant cardiac disease in the judgment of the investigator.
12. History of clinically significant electrocardiograms (ECG) abnormalities, or any of the following ECG abnormalities at screening or baseline:

    * PR greater than (>) 200 milliseconds (msec)
    * QRS complex >120 msec
    * Fridericia QT correction formula (QTcF) greater than (>) 450 msec
    * History of familial long QT syndrome or known family history of ventricular arrythmia.
    * Acute ischemic changes.
13. History or presence of mental illness evidenced as defined in the protocol.
14. Abnormal neurological condition or abnormal neurological examination at screening in judgment of investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Weekly-mean 24-hour Average Pain Score on the Numeric Rating Scale (NRS) at Week 15 | Baseline and at Week 15
  The NRS is an 11-point scale with scores ranging from 0 (no pain) to 10 (worst pain imaginable) for measuring participant self-reporting of pain intensity. A reduction in the score over time represents an improvement.

SECONDARY OUTCOMES:
Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) | Baseline up to Week 19
  The NPSI is a 12-items patient reported outcome (PRO) measure that contains 10 descriptors representing 5 dimensions of pain (burning pain, deep/pressing pain, paroxysmal pain, evoked pain, and paresthesia/dysesthesia), and 2 temporal items designed to assess pain duration and the number of pain paroxysms. Total score range for NPSI is 0-100, higher scores indicate more severity.
Change From Baseline in Brief Pain Inventory - Short Form (BPI-SF) Scale | Baseline up to Week 19
  The BPI-SF allows participants to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function using a 0 to 10 NRS. A higher score indicates more severity or more interference.
Change From Baseline in Weekly-mean 24-hour Average, Worst and Least Pain Score on the NRS | Baseline up to Week 19
  The NRS is an 11-point scale with scores ranging from 0 (no pain) to 10 (worst pain imaginable) for measuring participant self-reporting of pain intensity. A reduction in the score over time represents an improvement.
Proportion of Participants Achieving at least 30 Percent (%) and 50% Reduction From Baseline in the Weekly-mean 24-hour Average Pain Score on the NRS | Baseline up to Week 19
  The NRS is an 11-point scale with scores ranging from 0 (no pain) to 10 (worst pain imaginable) for measuring participant self-reporting of pain intensity. A reduction in the score over time represents an improvement.
Proportion of Participants with Treatment-emergent Adverse Events (TEAEs) and Their Severity | Baseline up to Week 19
Proportion of Participants With Adverse Events (AEs) Leading to Study Treatment Discontinuation and Adverse Events of Special Interest (AESI) and Serious Adverse Events (SAEs). | Baseline up to Week 19
Assessment of Diabetic Neuropathy using the Michigan Neuropathy Screening Instrument (MNSI) - Part B | Baseline up to Week 19
  The MNSI Part B consists of visual inspection of the feet and assessment of ankle reflexes, vibration sense, and monofilament testing. The measure is a score between 0 (normal) and 10 (most severe).
Assessment of Suicidal Ideation and Behavior using the Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline up to Week 19
  The C-SSRS is a semi-structured interview to assess the presence and severity of suicidal ideation and behavior.
Assessment of Withdrawal Symptoms After Termination of Study Treatment using the Study Medication Withdrawal Questionnaire Version 2 (SMWQ V2) | Baseline up to Week 19
  The SMWQ V2 is a 10-item patient-reported measure, where responses related to withdrawal symptoms are rated on 5-level Lickert scales between 0 (not at all) and 4 (very much).
Number of Participants With Clinically Significant Abnormal Lung Function Measured using Spirometry | Baseline up to Week 19
  Spirometry is a test that measures how much air can be breathed out in one forced breath. It is used to measure acute effects of study treatment on lung function. Spirometry testing will include measurement of forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), and FEV1/FVC.
Number of Participants With Clinically Significant Abnormality in Electrocardiogram (ECG) | Baseline up to Week 19
  An ECG is a test that records the electrical activity of the heart. It is used to measure acute effects of study treatment on heart function.
Number of Participants With Clinically Significant Abnormality in Blood and Urine Parameters | Baseline up to Week 19
  A variety of laboratory tests will be used to identify any clinically significant abnormalities.
Pharmacokinetics - Ctrough | At selected visits from baseline up to Week 16
  Pre-dose plasma concentration (Ctrough) of Δ9-THC, cannabidiol, cannabinol, 11-OH-THC, and 11-COOH-THC.
Pharmacokinetics - Cmax,ss | At selected visits from baseline up to Week 16
  Maximum observed plasma steady state concentration (Cmax,ss) for Δ9-THC, cannabidiol, cannabinol, 11-OH-THC, and 11-COOH-THC.
Pharmacokinetics - Tmax,ss | At selected visits from baseline up to Week 16
  Time to reach maximum observed plasma steady state concentration (Tmax,ss) for Δ9-THC, cannabidiol, cannabinol, 11-OH-THC, and 11-COOH-THC.
Pharmacokinetics - AUC | At selected visits from baseline up to Week 16
  Area under the concentration-time curve (AUC) for Δ9-THC, cannabidiol, cannabinol, 11-OH-THC, and 11-COOH-THC.
Proportion of Participants who Need Rescue Medication for the Treatment of DPNP | Baseline up to Week 19
Frequency of Rescue Medication Taken for the Treatment of DPNP | Baseline up to Week 19
Amount of Rescue Medication Taken for the Treatment of DPNP | Baseline up to Week 19
Time to First Intake of Rescue Medication Taken for the Treatment of DPNP | Baseline up to Week 19
Change From Baseline in Weekly-mean 24-hour Sleep Score Using the Daily Sleep Interference Scale (DSIS) | Baseline up to Week 19
  The DSIS diary consists of an 11-point Likert scale with which participants assess how pain has interfered with their sleep during the past 24 hours. On this scale a 0 indicates "pain does not interfere with sleep" and 10 indicates "pain completely interferes with sleep." A higher score indicates more inference of pain with sleep.
Change From Baseline in Sleep Score Using the Pain and Sleep Questionnaire-3 (PSQ-3) | Baseline up to Week 19
  The PSQ-3, also called Chronic Pain Sleep Inventory©, is a patient-reported 3-item index to assess the impact of chronic pain on sleep over the past 7 days. Each item is reported on a visual analog scale (VAS) between "never" and "always". The score ranges from 0 to 100.
Change From Baseline in Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) Profile Total Score | Baseline up to Week 19
  PROMIS-29 Profile v2.1 is a set of person-centered measures that evaluates and monitors physical, mental, and social health. PROMIS-29 Profile v2.1 consists of 7 domains with a total of 29 questions answered on Lickert scales.

CONTACTS AND LOCATIONS:
Overall Officials: Edith Dekel, Study Director — Syqe Medical Ltd.
Locations (38):
- Australia (5):
  - Innovate Clinical Research, Waitara, New South Wales
  - Western Sydney University NICM Health Research Institute (NICM HRI), Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Emeritus Research, Camberwell, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Czechia (4):
  - Rychnov nad Kneznou, Hradec Kralove, Rychnov nad Kněžnou, Hradec Kralove
  - Ostrava, Ostrava City, Ostrava, Ostrava City
  - Plzen, Plzen City, Pilsen, Plzen City
  - Prague, Praha 12, Prague, Prague
- Germany (11):
  - Heidelberg, Baden-Wuerttemberg, Heidelberg, Baden-Wurttemberg
  - Karlsruhe, Baden-Württemberg, Karlsruhe, Baden-Wurttemberg
  - Ulm, Baden-Württemberg, Ulm, Baden-Wurttemberg
  - Hamburg, Hamburg, Hamburg, Hamburg
  - Hannover, Lower Saxony, Hanover, Lower Saxony
  - Schwerin, Mecklenburg, Schwerin, Mecklenburg
  - Reinfeld, Schleswig-Holstein, Reinfeld, Schleswig-Holstein
  - Berlin, Berlin 4010, Berlin, State of Berlin
  - Berlin, Berlin, Berlin, State of Berlin
  - Klinische Forschung Dresden GmbH, Dresden
  - Klinische Forschung Schwerin GmbH, Schwerin
- Israel (8):
  - The Edith Wolfson Medical Center, Holon, Tel Aviv
  - Sheba Medical center Hospital, Ramat Gan, Tel Aviv
  - Barzilai Medical center, Ashkelon
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Beilinson hospital/ Petach Tikva, Petah Tikva
  - Ziv Medical Center, Safed
- Poland (10):
  - Swidnica, Dolnoslaskie, Swidnica, Lower Silesian Voivodeship
  - Sochaczew, Mazowieckie, Sochaczew, Masovian Voivodeship
  - Warszawa, Mazowieckie 7011, Warsaw, Masovian Voivodeship
  - Warszawa, Mazowieckie, Warsaw, Masovian Voivodeship
  - Warszawa, Mazowieckie 7010, Warsaw, Masovian Voivodeship
  - Katowice, Silesia, Katowice, Silesian Voivodeship
  - Katowice, Śląsk, Katowice, Silesian Voivodeship
  - Centrum Medyczne NEUROMED, Bydgoszcz
  - Centrum Medyczne Pratia Chojnice, Chojnice
  - Osrodek Badan Klinicznych Neuro-Medic Clinic, Katowice

IPD SHARING:
Plan to Share IPD: Undecided